CLINICAL TRIAL: NCT04740502
Title: Surgical Approach and Outcomes in Patients With Primary Hyperparathyroidism and Unclear Preoperative Localisation Studies
Brief Title: Surgical Outcomes in Patients With Primary Hyperparathyroidism and Unclear Preoperative Localisation Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Assistant Professor, University of Cagliari
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHP-DISC
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concordant preoperative studies (Other): Patients with concordant neck ultrasound and MIBI scan
  Interventions: Procedure: Parahtyroidectomy
- Unclear preoperative studies (Other): Patients with discordant or negative neck ultrasound and MIBI scan
  Interventions: Procedure: Parahtyroidectomy

INTERVENTIONS:
Procedure: Parahtyroidectomy — Parathyroidectomy

SUMMARY:
Although some surgeons still consider bilateral neck exploration as the best approach for primary hyperparathyroidism, nowadays most of them perceive the mini-invasive parathyroidectomy (MIP) as the best option for patients with concordant preoperative studies. Nevertheless, the consensus is heterogeneous for patients with unclear localisation studies, with some surgeons deeming BNE as mandatory and others suggesting that a mini-invasive approach is still possible if combined with IOPTH monitoring. In our research, we focused on patients with unclear preoperative localisation studies, to better understand the factors that can determine discordant or negative results between US and MIBI scan, in order to choose the best surgical approach and to evaluate the outcomes in this kind of patients.

DETAILED DESCRIPTION:
This is an unicentric, retrospective study on patients who underwent surgery for PHP from January 2004 to June 2020 at our Department of General and Endocrine surgery, which is a tertiary referral centre for parathyroid disease. Ethical approval was released from our Local Independent Ethical Committee. Patients involved in the study subjects gave informed consent to the work.

In our study, we included only patients who underwent both US and MIBI preoperatively. The exclusion criteria were the association of total or partial thyroidectomy planned preoperatively for thyroid disease, reoperative surgery for persistent or recurrent PHP, and incomplete data or follow-up.

The primary aims of this study were:

* To identify predictive factors of unclear preoperative localisation studies.
* To evaluate if a mini-invasive approach is feasible in this kind of patients, considering the incidence of persistent PHP as the main outcome.

The secondary outcomes were:

* To assess the role of IOPTH assay in patients with unclear localisation studies.
* To evaluate the accuracy of preoperative localisation studies in our series, particularly in patients with discordant or negative US and MIBI scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hyperparathyroidism

Exclusion Criteria:

* Patients with concomitant thyroid disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Surgical failure | 6 months
  Incidence of persistent hyperparathyroidism

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Policlinico di Monserrato, Monserrato, Cagliari
  - Policlinico di Monserrato, Monserrato, CA

IPD SHARING:
Plan to Share IPD: Undecided